CLINICAL TRIAL: NCT03907696
Title: Reducing Stigma Towards Psychiatry Among Medical Students: a Multicenter Controlled Trial
Brief Title: Reducing Stigma Towards Psychiatry Among Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Raz Gross, Raz Gross, MD, MPH, program director, Psychiatry, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 4716-17-SMC
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Stigma, Social
MeSH Terms: conditions — Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): The intervention arm participate in an educational program that aimed at reducing stigma
  Interventions: Other: Anti-stigma interventions curriculum
- control (No Intervention): regular curriculum with no addition educational contents

INTERVENTIONS:
Other: Anti-stigma interventions curriculum — educational curriculum aimed at reducing stigma
  Arms: Intervention

SUMMARY:
This study examines the effect of including a novel Anti-stigma Intervention Curriculum (ASIC) during a clinical rotation in psychiatry during medical school. It addresses stigma in medical students' perceptions of psychiatric patients, psychiatric illnesses and treatments, and the knowledge base of psychiatry in clinical practice.

Medical students from eight hospitals were divided into intervention (one hospital, n=57) and control (seven hospitals, n=163) arms at the beginning of a 6-week psychiatry rotation throughout one academic year (2017/18). The students completed the Attitudes to Psychiatry scale (ATP-30) and the Attitudes toward Mental Illness scale (AMI) at rotation onset and conclusion. The ASIC was designed to target prejudices and stigma by direct informal encounters with people with severe mental illness (SMI) during periods of remission and recovery. Supervised small group discussions followed those encounters in order to facilitate processing of thoughts and emotions that ensued, and to discuss salient topics, including psychiatric care, evidence-based medicine in psychiatry, and the neuroscientific underpinnings of clinical psychiatry.

DETAILED DESCRIPTION:
Design and participants- This study used a controlled trial design. The study population consisted of medical students during their six-week psychiatry clerkship. The study was conducted between November 2017 and July 2018 in eight academic hospitals in central Israel. There were 16 groups of students.

The intervention arm included 3 groups of students (n=57) at a single general hospital, and the control group was comprised of 13 groups of students (n=163) from six psychiatric hospitals (n=139) and one general hospital (n=24). All students were informed that the purpose of the study was to explore their attitudes about people with mental illness and about psychiatry in general at the beginning (baseline) and at the end (endpoint) of their rotation. The participants were assured that their responses would remain confidential, and that they would not influence their rotation grade.

Procedure - The intervention and control groups received the same lecture and practical training components. Topics covered in the lectures included psychopathology, psychopharmacological treatment, psychotherapy, and forensic psychiatry. Practical training included participation in inpatient rounds, visits at outpatient clinics and consultation-liaison services, and seminars consisting of patient interviews and discussions of clinical cases. All students were placed in a psychiatric ward, under the supervision and responsibility of psychiatric residents and senior psychiatrists. Each ward had a range of 4 to 7 students assigned to it. During the rotation, students assumed supervised clinical responsibility for at least one clinical case. Although all students were exposed to a variety of patients in different clinical scenarios, they were exposed mostly to acutely ill inpatients.

Study intervention The Anti-Stigma Interventions Curriculum (ASIC) component that was added to the intervention group was designed to target stigma towards psychiatric patients, psychiatric treatment, and the knowledge base of clinical practice in psychiatry. A first part, aimed at reducing stigma towards psychiatric patients, consisted of two forms of direct encounters with individuals with serious mental illness (SMI) in recovery or rehabilitation: 1) A two-hour panel of three people who shared their personal stories as consumers of mental health services, followed by an open discussion with the students; and 2) A visit to a rehabilitation center, which included direct contact with the consumers. The emphasis in both of those encounters was on exposing students to the competence and strengths of the individuals, rather than to the symptoms and signs of their underlying illnesses. The second part, which was designed to target stigma towards psychiatric treatment and the knowledge base of clinical practice in psychiatry, included small group discussions (20 minutes each) on the efficacy of different treatments, the clinical utility of admission to inpatient wards, evidence-based medicine in psychiatry, and the biological pathways underpinning psychiatric disorders.

The study was conducted after receiving Helsinki ethics committee approval for a multicenter study from the University of Tel Aviv Institutional Review Board. Because the ethics committee approval was contingent on personal information being de-identified, the investigators only used aggregate, unpaired pre- and post-rotation data.

Study evaluations Participants completed one socio-demographic and two self-report questionnaires, the Attitudes to Psychiatry (ATP-30)22, and the Attitudes to Mental Illness (AMI)7, which were administrated through a secured online server (SurveyMonkey®). The ATP-30 consists of 30 items, and it measures medical students' attitudes towards eight different attitudinal domains: 1) Psychiatric patients; 2) Psychiatric illness; 3) Psychiatric treatment; 4) Psychiatric institutions; 5) Psychiatric knowledge base in clinical practice; 6) Psychiatric education; 7) Psychiatry as a career choice; and 8) Psychiatrists. The AMI consists of 20 items, and it measures medical students' attitudes to mental illnesses and, more specifically, towards their causes, treatments, and impact on individuals and society. Each item in both questionnaires is rated on a 5-point Likert scale ranging from strongly agree to strongly disagree. Some items are negatively phrased in order to minimize the likelihood of social desirability bias, and higher composite scores indicate more favorable attitudes (less stigma) toward mental illness. Both ATP-30 and AMI have been shown to have good psychometric properties, and both have been translated into many languages and used in many countries worldwide.7,22

ELIGIBILITY:
Inclusion Criteria:

- All medical students in psychiatric rotation during the academic year of 2017-2018 affiliated to Tel Aviv University

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Attitude toward psychiatry (ATP) scale | 6 weeks (psychiatric rotation)
  scale that measure stigma among medical students. 30 statements, scale of 1 (strongly disagree) to 5 (strongly agree). Minimum score: 30; maximum score: 150; Higher scores indicate less stigma.
Attitude toward mental illness (AMI) scale | 6 weeks (psychiatric rotation)
  scale that measure stigma among medical students. 30 statements, scale of 1 (strongly disagree) to 5 (strongly agree). Minimum score: 20; maximum score: 100. Higher scores indicate less stigma.

CONTACTS AND LOCATIONS:
Overall Officials: Doron Amsalem, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Doron Amsalem, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
Individual participant data is not available for other researchers

REFERENCES:
- [Derived] Amsalem D, Gothelf D, Dorman A, Goren Y, Tene O, Shelef A, Horowitz I, Dunsky LL, Rogev E, Klein EH, Mekori-Domachevsky E, Fischel T, Levkovitz Y, Martin A, Gross R. Reducing Stigma Toward Psychiatry Among Medical Students: A Multicenter Controlled Trial. Prim Care Companion CNS Disord. 2020 Feb 27;22(2):19m02527. doi: 10.4088/PCC.19m02527. PMID 32135042